CLINICAL TRIAL: NCT02822859
Title: A Comparison of Three Nebulizers for Standard Clinical and Research Use in Methacholine Challenge Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, MD, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCH NEB-1
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wright (Active Comparator): Methacholine challenge performed using the Wright nebulizer
  Interventions: Device: Wright nebulizer
- Bennett-Twin (Active Comparator): Methacholine challenge performed using the Bennett-Twin nebulizer
  Interventions: Device: Bennett-Twin nebulizer
- Aeroneb Solo (Active Comparator): Methacholine challenge performed using the Aeroneb Solo nebulizer
  Interventions: Device: Aeroneb Solo

INTERVENTIONS:
Device: Wright nebulizer — Roxon Medi-Tech, Montreal, QC, Canada
  Arms: Wright
Device: Bennett-Twin nebulizer — Puritan Bennett Corp., Carlsbad, CA, USA
  Arms: Bennett-Twin
Device: Aeroneb Solo — Aerogen Ltd., Galway, Ireland
  Arms: Aeroneb Solo

SUMMARY:
The study will assess three different nebulizers for use in methacholine challenge testing in order to determine if the Aeroneb Solo would make a suitable replacement for the long-used and now obsolete Wright and Bennett-Twin nebulizers. Results from each device will be compared to evaluate whether current guidelines for the methacholine challenge should be updated for superior standardization.

DETAILED DESCRIPTION:
Sixty asthmatics (20 at each testing site: University of Saskatchewan, McMaster University, Laval University) will be recruited to undergo this randomized, triple cross-over study. Three nebulizers will be tested, the Wright, the Bennett-Twin and the new Aeroneb Solo.

Breakdown of study procedure: Participants will undergo three (potentially four) methacholine challenges, one with each nebulizer in randomized order. An additional methacholine challenge may be performed for screening purposes if the participant has not undergone methacholine challenge testing in one of the participating labs in the previous 6 months. The screening challenge will be performed with the standard nebulizer used at the given testing site (i.e. the Wright or the Bennett-Twin).

The methacholine challenges performed with the Wright and Bennett-Twin nebulizers will follow the two-minute tidal breathing protocol as outlined in the 1999 American Thoracic Society Guidelines for Methacholine Challenge Testing. The testing protocol used with the Aeroneb solo will be identical save for a 1 min inhalation period instead of 2 min. Each challenge will be stopped when a participant's forced expiratory volume in 1 second (FEV1) drops at least 20%. This will allow for the determination of the participant's PC20 (provocative concentration of methacholine causing a 20% fall in FEV1), which will subsequently be converted to a PD20 (provocative dose) value. A minimum 24-hour washout period between challenges will be enforced.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older
* Stable asthma
* Baseline methacholine PC20 less than or equal to 16mg/mL
* Baseline lung function greater than 65% predicted

Exclusion Criteria:

* Use of long-acting bronchodilators within 30 days of Visit 1
* Pregnant or nursing
* Cardiovascular problems
* Respiratory illness within 4 weeks of Visit 1
* Allergen-induced asthma exacerbation within 4 weeks of Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
airway responsiveness to methacholine (methacholine pd20) | Two weeks
  methacholine pd20 data will be compared between nebulizers (Wright, Bennett and Solo). Methacholine PD20 data generated with the Wright nebulizer will serve as the comparator for the methacholine pd20 generated with the Bennett and the Solo nebulizers.

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Asthma Research Lab - University of Saskatchewan, Saskatoon, Saskatchewan
  - Laval University, Québec

IPD SHARING:
Plan to Share IPD: Yes
Journal Publication